CLINICAL TRIAL: NCT03115294
Title: Digital Image Correlation in Right Ventricular Evaluation in Cardiac Surgery
Brief Title: Digital Image Correlation in Right Ventricular Evaluation
Acronym: CardiomeDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other)
Responsible Party: Principal Investigator, Jari Laurikka, Professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: R16045
Record Dates: First submitted 2017-03-08; First posted 2017-04-14 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Heart Ventricles
MeSH Terms: interventions — Theophylline

STUDY DESIGN:
Intervention Model Description: Patients undergo medication intervention (w/intravenous theophylline) and ventilator volume adjustements, and serial ventricular function parameters are compared (pre-and post-intervention measurements).
Masking Description: video analysts do not get information of the clinical data or procedure phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients undergo procedure with stepwise measurements and ventilator + volume adjustment + iv theophylline Myocardial movement recording using videoscanning
  Interventions: Drug: Theophylline; Procedure: Ventilator positive end expiratory pressure adjustment; Device: Videorecording

INTERVENTIONS:
Drug: Theophylline — iv injection
Procedure: Ventilator positive end expiratory pressure adjustment — Positive end-expiratory pressure variation
Device: Videorecording — Myocardial movement videorecording

SUMMARY:
Observational study of patients undergoing open heart surgery. During the procedure video clips of right heart are stored and compared to trans-oesophageal ultrasound recordings and ECG recordings.

DETAILED DESCRIPTION:
Observational study of patients undergoing open heart surgery. During the procedure video clips of right heart are stored and compared to trans-oesophageal ultrasound recordings and ECG recordings. Right heart volume status and function is controlled and induced with theophylline and ventilator regulated positive end-expiratory pressure recordings.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery, patient acceptance and informed consent, age 75 or more

Exclusion Criteria:

* patient refusal, psychiatric disorder or intoxication, irrepairable coronary artery disease, epilepsy or active neurological condition, active tbc or other contagious infection.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Heart ventricle function | Within the operation
  Changes in heart ventricle contraction status

OTHER OUTCOMES:
ECG | Within the operation
  Simultaneous ECG recording and analysis during outcome 4 measurements
Transesophageal ultrasound | Within the operation
  Myocardial contraction range during video-clip
Cardiac output | Within the operation
  Measurement of cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Jari Laurikka, MD,PhD, Principal Investigator — Professor, Cardio-thoracic Surgery
Locations (1):
- Tampere University Hospital, Heart Center, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No
non-identifiable data to Tampere University of Technology research group

REFERENCES:
- [Result] Soltani A, Lahti J, Jarvela K, Laurikka J, Kuokkala VT, Hokka M. Characterization of the anisotropic deformation of the right ventricle during open heart surgery. Comput Methods Biomech Biomed Engin. 2020 Feb;23(3):103-113. doi: 10.1080/10255842.2019.1703133. Epub 2019 Dec 17. PMID 31847587
- [Result] Soltani A, Lahti J, Jarvela K, Curtze S, Laurikka J, Hokka M, Kuokkala VT. An Optical Method for the In-Vivo Characterization of the Biomechanical Response of the Right Ventricle. Sci Rep. 2018 May 1;8(1):6831. doi: 10.1038/s41598-018-25223-z. PMID 29717224